CLINICAL TRIAL: NCT01457118
Title: An Open-Label, Multicenter, Extension Study of NKTR-102 in Subjects Previously Enrolled in NKTR-102 Studies
Brief Title: An Extension Study of NKTR-102 in Cancer Patients Previously Enrolled in NKTR-102 Studies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-PIR-09
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Malignant Solid Tumor
Keywords: Open Label multicenter extension study advanced solid tumors
MeSH Terms: interventions — etirinotecan pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NKTR-102 (Experimental)
  Interventions: Drug: NKTR-102 145 mg/m2; Drug: NKTR-102 120 mg/m2; Drug: NKTR-102 95 mg/m2; Drug: NKTR-102 50 mg/m2

INTERVENTIONS:
Drug: NKTR-102 145 mg/m2 — A 90 minute IV infusion of 145 mg/m2 or less of NKTR-102 on Day 1 of each 21-day treatment cycle.
Drug: NKTR-102 120 mg/m2 — A 90 minute IV infusion of 120 mg/m2 or less of NKTR-102 on Day 1 of each 21-day treatment cycle.
Drug: NKTR-102 95 mg/m2 — A 90 minute IV infusion of 95 mg/m2 or less of NKTR-102 on Day 1 of each 21-day treatment cycle.
Drug: NKTR-102 50 mg/m2 — A 90 minute IV infusion of 50 mg/m2 or less of NKTR-102 on Day 1 of each 21-day treatment cycle.

SUMMARY:
The study objective of this open label, multicenter study is to provide access to NKTR-102 treatment to subjects previously enrolled in a NKTR-102 study who are without signs of disease progression since receiving NKTR-102.

In addition the study will evaluate the safety of continued exposure to NKTR-102, observe disease status and survival status in subjects receiving NKTR-102, and evaluate the efficacy of NKTR-102 in subjects with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion:

1. Received prior treatment with NKTR-102
2. Free of disease progression since receiving NKTR-102
3. Adequate bone marrow and organ function
4. Treatment with NKTR-102 in the extension study to begin within 8 weeks after receipt of their of last dose of NKTR-102
5. Agree to use adequate contraception

Exclusion:

1. Treatment with other anti-cancer therapy between the last dose of NKTR-102 in the prior study and before first dose of NKTR-102 in the extension study
2. A toxicity that requires a 3rd dose reduction after taking NKTR-102 or are scheduled to receive a dose < 70 mg/m2 upon entry into this study
3. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (7):
- United States (5):
  - Investigator Site - Los Angeles, Los Angeles, California
  - Investigator Site - San Francisco, San Francisco, California
  - Investigator Site - Whittier, Whittier, California
  - Investigator Site - Minneapolis, Minneapolis, Minnesota
  - Investigator Site - Cleveland, Cleveland, Ohio
- Belgium (2):
  - Investigator Site - Bruxelles, Brussels
  - Investigator Site - Liege, Liège

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were assessed for eligibility following completion of NKTR-102 treatment on a prior NKTR-102 clinical study. The trials from which the subjects were previously enrolled in are listed below.
  NCT00856375 - 1 patient NCT00806156 - 1 patient NCT01492101 - 1 patient NCT00802945 - 2 patients NCT01976143 - 10 patients NCT01991678 - 12 patients
Groups:
- 145 mg/m2: NKTR-102: A 90 minute IV infusion of 145 mg/m2
- 120 mg/m2: NKTR-102: A 90 minute IV infusion of 120 mg/m2
- 95 mg/m2: NKTR-102: A 90 minute IV infusion of 95 mg/m2
- 50 mg/m2: NKTR-102: A 90 minute IV infusion of 50 mg/m2
Period: Overall Study
Arm/Group | 145 mg/m2 | 120 mg/m2 | 95 mg/m2 | 50 mg/m2
Started | 20 | 4 | 1 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 20 | 4 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 1
Not completed — Clinical Progression | 0 | 1 | 0 | 1
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Progressive Disease by RECIST | 12 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 145 mg/m2 | 120 mg/m2 | 95 mg/m2 | 50 mg/m2 | Total
Number analyzed (Participants) | 20 | 4 | 1 | 2 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (9.92) | 63.0 (9.98) | 44.0 (NA) — There is only one participant | 53.5 (3.54) | 56.0 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 2 | 1 | 1 | 17
  Male | 7 | 2 | 0 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 2 | 5
  Not Hispanic or Latino | 17 | 3 | 1 | 0 | 21
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 14 | 4 | 0 | 2 | 20
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Primary Tumor Diagnosis [Count of Participants; unit: Participants]
  Breast | 3 | 0 | 1 | 0 | 4
  Colorectal | 8 | 2 | 0 | 0 | 10
  Liver | 0 | 1 | 0 | 2 | 3
  Lung | 1 | 0 | 0 | 0 | 1
  Other | 5 | 0 | 0 | 0 | 5
  Ovary | 1 | 1 | 0 | 0 | 2
  Pancreas | 2 | 0 | 0 | 0 | 2
Stage at Original NKTR-102 Study Enrollment [Count of Participants; unit: Participants]
  I | 2 | 1 | 0 | 2 | 5
  II | 3 | 1 | 0 | 0 | 4
  IIA | 0 | 0 | 1 | 0 | 1
  III | 4 | 1 | 0 | 0 | 5
  IV | 7 | 0 | 0 | 0 | 7
  Unknown | 4 | 1 | 0 | 0 | 5
Time Since Initial Diagnosis to Original NKTR-102 Study [Mean (Standard Deviation); unit: years] | 5.936 (5.3536) | 5.040 (1.2142) | 15.780 (NA) — There is only one participant | 3.450 (0.0707) | 5.984 (5.0437)
Treatment Duration in Original NKTR-102 Study [Mean (Standard Deviation); unit: days] | 56.6 (125.67) | 141.5 (179.04) | 1008.0 (NA) — There is only one participant | 21.0 (0.00) | 101.7 (221.68)
Time Since Metastatic Diagnosis to Original NKTR-102 Study [Mean (Standard Deviation); unit: days] — Population: The number analyzed differs from overall as not all patients reached metastatic diagnosis
  days
    number analyzed (Participants) | 18 | 4 | 1 | 1 | 24
    (all) | 3.666 (2.3677) | 2.733 (1.3546) | 3.660 (NA) — There is only one patient | 0.000 (NA) — There is only one patient | 3.357 (2.2403)

OUTCOME MEASURES:

1. Primary Outcome: Length of Exposure to NKTR-102
Description: To provide access to NKTR-102 to subjects who previously received NKTR-102 in a clinical trial and were without signs of disease progression since receiving NKTR-102.
Time Frame: Screening, Every 21 day cycle of treatment and Quarterly Follow-up
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 145 mg/m2 | 120 mg/m2 | 95 mg/m2 | 50 mg/m2
Number analyzed (Participants) | 20 | 4 | 1 | 2
days | 139.0 (126.19) | 33.0 (14.07) | 126.0 (NA) — There is only one participant | 21.0 (0.00)

2. Secondary Outcome: Adverse Events
Description: To evaluate the safety of continued exposure to NKTR-102.
Time Frame: Screening, Every 21 day cycle of treatment and Quarterly Follow-up
Measure: Number; unit: # of events
Arm/Group | 145 mg/m2 | 120 mg/m2 | 95 mg/m2 | 50 mg/m2
Number analyzed (Participants) | 20 | 4 | 1 | 2
# of events
  # of Subjects with Anemia | 3 | 1 | 0 | 0
  # of Subjects with Neutropenia | 3 | 0 | 0 | 0
  # of Subjects with Leukopenia | 1 | 0 | 0 | 0
  # of Subjects with Tachycardia | 1 | 0 | 0 | 0
  # of Subjects with Vision Blurred | 3 | 1 | 0 | 0
  # of Subjects with Photophobia | 1 | 0 | 0 | 0
  # of Subjects with Diarrhea | 11 | 3 | 0 | 0
  # of Subjects with Nausea | 6 | 0 | 0 | 0
  # of Subjects with Vomiting | 4 | 2 | 0 | 0
  # of Subjects with Constipation | 4 | 1 | 0 | 0
  # of Subjects with Abdominal Pain | 2 | 1 | 0 | 1
  # of Subjects with Dyspepsia | 2 | 0 | 0 | 0
  # of Subjects with Upper Abdominal Pain | 1 | 0 | 0 | 0
  # of Subjects with Ascites | 0 | 0 | 0 | 1
  # of Subjects with Dry Mouth | 0 | 1 | 0 | 0
  # of Subjects with Hypoaesthesia Oral | 1 | 0 | 0 | 0
  # of Subjects with Mouth Ulceration | 1 | 0 | 0 | 0
  # of Subjects with Stomatitis | 1 | 0 | 0 | 0
  # of Subjects with Fatigue | 6 | 1 | 0 | 1
  # of Subjects with Oedema Peripheral | 2 | 0 | 0 | 0
  # of Subjects with Non-Cardiac Chest Pain | 1 | 0 | 0 | 0
  # of Subjects with Pyrexia | 1 | 0 | 0 | 0
  # of Subjects with Urinary Tract Infections | 3 | 0 | 0 | 0
  # of Subjects with Gastroenteritis | 1 | 1 | 0 | 0
  # of Subjects with Influenza | 0 | 1 | 1 | 0
  # of Subjects with Abdominal Infection | 0 | 1 | 0 | 0
  # of Subjects with Gingival Infection | 1 | 0 | 0 | 0
  # of Subjects with Herpex Simplex Encephalitis | 0 | 0 | 0 | 1
  # of Subjects with Weight Decreased | 5 | 0 | 0 | 0
  # of Subjects with Neutrophil Count Decreased | 1 | 1 | 1 | 0
  # of Subjects with Aspartate Aminostransferase | 1 | 1 | 0 | 0
  # of Subjects with White blood cell count decreased | 1 | 1 | 0 | 0
  # of Subjects with Activated partial thromboplastin time prolonged | 0 | 1 | 0 | 0
  # of Subjects with Alanine Aminotransferase Increased | 1 | 0 | 0 | 0
  # of Subjects with Blood bilirubin increased | 1 | 0 | 0 | 0
  # of Subjects with Blood creatine increased | 1 | 0 | 0 | 0
  # of Subjects with Liver Function Test abnormal | 1 | 0 | 0 | 0
  # of Subjects with Prothrombin time prolonged | 1 | 0 | 0 | 0
  # of Subjects with decreased appetite | 4 | 0 | 1 | 1
  # of Subjects with hypoalbuminemia | 3 | 1 | 0 | 0
  # of Subjects with hypokalemia | 2 | 1 | 0 | 0
  # of Subjects with hypoglycemia | 1 | 1 | 0 | 0
  # of Subjects with hyponatremia | 2 | 0 | 0 | 0
  # of Subjects with dehydration | 0 | 1 | 0 | 0
  # of Subjects with Hyperglycemia | 1 | 0 | 0 | 0
  # of Subjects with Hypocalcemia | 1 | 0 | 0 | 0
  # of Subjects with Hypomagnesemia | 1 | 0 | 0 | 0
  # of Subjects with Hypophosphatemia | 1 | 0 | 0 | 0
  # of Subjects with Back Pain | 1 | 0 | 0 | 0
  # of Subjects with Flank Pain | 1 | 0 | 0 | 0
  # of Subjects with Muscular Weakness | 0 | 1 | 0 | 0
  # of Subjects with Musculoskeletal Pain | 0 | 1 | 0 | 0
  # of Subjects with Appendix Cancer | 1 | 0 | 0 | 0
  # of Subjects with Cancer Pain | 1 | 0 | 0 | 0
  # of Subjects with Aphonia | 1 | 0 | 0 | 0
  # of Subjects with Dyasgeusia | 1 | 0 | 0 | 0
  # of Subjects with Hypoaesthsia | 1 | 0 | 0 | 0
  # of Subjects with Depressed Mood | 1 | 0 | 0 | 0
  # of Subjects with Insomnia | 0 | 0 | 0 | 1
  # of Subjects with Proteinuria | 1 | 0 | 0 | 0
  # of Subjects with Renal Failure Acute | 1 | 0 | 0 | 0
  # of Subjects with Vaginal Hemorrhage | 1 | 0 | 0 | 0
  # of Subjects with Oropharyngeal Pain | 2 | 1 | 0 | 0
  # of Subjects with Cough | 1 | 0 | 0 | 0
  # of Subjects with Dsypnoea | 1 | 0 | 0 | 0
  # of Subjects with Epistaxis | 1 | 0 | 0 | 0
  # of Subjects with Hypoxis | 1 | 0 | 0 | 0
  # of Subjects with Pneumothorax | 1 | 0 | 0 | 0
  # of Subjects with Productive Cough | 1 | 0 | 0 | 0
  # of Subjects with Pulmonary Embolism | 1 | 0 | 0 | 0
  # of Subjects with Decubitus Ulcer | 2 | 0 | 0 | 0
  # of Subjects with Pruritus | 1 | 0 | 0 | 1
  # of Subjects with Rash | 2 | 0 | 0 | 0
  # of Subjects with Alopecia | 1 | 0 | 0 | 0
  # of Subjects with Hypotension | 1 | 0 | 0 | 0
  # of Subjects with Pelvic Venous Thrombosis | 1 | 0 | 0 | 0
  Number of Subjects with at least one TEAE | 20 | 4 | 1 | 2
  # of Subjects with Peritonitis Bacterial | 0 | 1 | 0 | 0

3. Secondary Outcome: Disease Status
Description: To observe disease status and survival status in subjects receiving NKTR-102.
Time Frame: Screening, Every 21 day cycle of treatment and Quarterly Follow-up
Population: Four participants including the one in Group 4 had to discontinue treatment prior to measuring this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | 145 mg/m2 | 120 mg/m2 | 95 mg/m2 | 50 mg/m2
Number analyzed (Participants) | 18 | 4 | 1 | 0
Participants
  Stable Disease (SD) | 10 | 1 | 0 | 0
  Progressive Disease (PD) | 8 | 3 | 1 | 0

4. Secondary Outcome: Efficacy of NKTR-102
Description: To evaluate the efficacy of NKTR-102 in subjects with advanced or metastatic solid tumors.
Time Frame: Screening, Every 21 day cycle of treatment and Quarterly Follow-up
Population: Four participants including the one in Group 4 had to discontinue treatment prior to this outcome being measured.
Measure: Number; unit: participants
Arm/Group | 145 mg/m2 | 120 mg/m2 | 95 mg/m2 | 50 mg/m2
Number analyzed (Participants) | 18 | 4 | 1 | 0
participants
  # of Participants who achieved Complete Response (CR) | 0 | 0 | 0 |
  # of Participants who achieved Partial Response (PR) | 0 | 0 | 0 |

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study approximately 6 years
Arm/Group | 145 mg/m2 | 120 mg/m2 | 95 mg/m2 | 50 mg/m2
All-Cause Mortality (participants affected / at risk) | 16/20 | 3/4 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 5/20 | 1/4 | 0/1 | 1/2
Other Adverse Events (participants affected / at risk) | 20/20 | 4/4 | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 145 mg/m2 (N=20) | 120 mg/m2 (N=4) | 95 mg/m2 (N=1) | 50 mg/m2 (N=2)
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal Infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Herpex simplex encephalitis (Infections and infestations) | 0 | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Appendix Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Total Number of TESAEs (General disorders) | 5 (10) | 1 (3) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 145 mg/m2 (N=20) | 120 mg/m2 (N=4) | 95 mg/m2 (N=1) | 50 mg/m2 (N=2)
# of subjects with Anemia (Cardiac disorders) | 3 | 1 | 0 | 0
# of subjects with Neutropenia (Immune system disorders) | 3 | 0 | 0 | 0
# of subjects with Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
# of subjects with Vision Blurred (Eye disorders) | 3 | 1 | 0 | 0
# of subjects with Photophobia (General disorders) | 1 | 0 | 0 | 0
# of subjects with Diarrhea (Gastrointestinal disorders) | 11 | 3 | 0 | 0
# of subjects with Nausea (Gastrointestinal disorders) | 6 | 0 | 0 | 0
# of subjects with Vomiting (Gastrointestinal disorders) | 4 | 2 | 0 | 0
# of subjects with Constipation (Gastrointestinal disorders) | 4 | 1 | 0 | 0
# of subjects with Abdominal Pain (General disorders) | 2 | 1 | 0 | 1
# of subjects with Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
# of subjects with Upper Abdominal Pain (General disorders) | 1 | 0 | 0 | 0
# of subjects with Ascites (Hepatobiliary disorders) | 0 | 0 | 0 | 1
# of subjects with Dry Mouth (General disorders) | 0 | 1 | 0 | 0
# of subjects with Hypoesthesia Oral (Nervous system disorders) | 1 | 0 | 0 | 0
# of subjects with Mouth Ulceration (Infections and infestations) | 1 | 0 | 0 | 0
# of subjects with Stomatitis (Infections and infestations) | 1 | 0 | 0 | 0
# of subjects with Fatigue (General disorders) | 6 | 1 | 0 | 1
# of subjects with Oedema Peripheral (Cardiac disorders) | 2 | 0 | 0 | 0
# of subjects with Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0
# of subjects with Pyrexia (General disorders) | 1 | 0 | 0 | 0
# of subjects with Urinary Tract Infections (Infections and infestations) | 3 | 0 | 0 | 0
# of subjects with Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0
# of subjects with Influenza (Infections and infestations) | 0 | 1 | 1 | 0
# of subjects with Abdominal Infection (Infections and infestations) | 0 | 1 | 0 | 0
# of subjects with Gingival Infection (Infections and infestations) | 1 | 0 | 0 | 0
# of subjects with Herpes Simplex Encephalitis (Infections and infestations) | 0 | 0 | 0 | 1
# of subjects with Weight Decreased (General disorders) | 5 | 0 | 0 | 0
# of subjects with Neutrophil Count Decreased (Immune system disorders) | 1 | 1 | 1 | 0
# of subjects with Aspartate Aminotransferase Increased (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
# of subjects with White Blood Cell count decreased (Immune system disorders) | 1 | 1 | 0 | 0
# of subjects with Activated Partial Thromboplastin Time Prolonged (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
# of subjects with Alanine Aminotransferase Increased (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
# of subjects with Blood Bilirubin Increased (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
# of subjects with Liver Function Test Abnormal (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
# of subjects with Prothrombin Time Prolonged (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
# of subjects with Decreased Appetite (General disorders) | 4 | 0 | 1 | 1
# of subjects with Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0
# of subjects with Hypokalemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
# of subjects with Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
# of subjects with Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
# of subjects with Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
# of subjects with Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
# of subjects with Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
# of subjects with Hypomagenesemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
# of subjects with Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
# of subjects with Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
# of subjects with Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
# of subjects with Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
# of subjects with Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
# of subjects with Appendix Pain (General disorders) | 1 | 0 | 0 | 0
# of subjects with Cancer Pain (General disorders) | 1 | 0 | 0 | 0
# of subjects with Aphonia (General disorders) | 1 | 0 | 0 | 0
# of subjects with Dysgeusia (General disorders) | 1 | 0 | 0 | 0
# of subjects with Hypoesthesia (General disorders) | 1 | 0 | 0 | 0
# of subjects with Depressed Mood (Psychiatric disorders) | 1 | 0 | 0 | 0
# of subjects with Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
# of subjects with Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
# of subjects with Acute Renal Failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
# of subjects with Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
# of subjects with Oropharyngeal Pain (General disorders) | 2 | 1 | 0 | 0
# of subjects with Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
# of subjects with Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
# of subjects with Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
# of subjects with Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
# of subjects with Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
# of subjects with Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
# of subjects with Pulmonary Embolism (Vascular disorders) | 1 | 0 | 0 | 0
# of subjects with Decubitus Ulcer (Infections and infestations) | 2 | 0 | 0 | 0
# of subjects with Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
# of subjects with Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
# of subjects with Alopecia (General disorders) | 1 | 0 | 0 | 0
# of subjects with Hypotension (Cardiac disorders) | 1 | 0 | 0 | 0
# of subjects with Pelvic Venous Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
# of subjects with Peritonitis Bacterial (Infections and infestations) | 1 | 0 | 0 | 0
# of subjects with Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
# of subjects with Blood Creatine Increased (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.

DOCUMENTS (2):
  • Study Protocol (2016-01-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT01457118/Prot_000.pdf
  • Statistical Analysis Plan (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT01457118/SAP_001.pdf